CLINICAL TRIAL: NCT03527433
Title: A Randomized, Controlled Trial Comparing Wound COmplications in Elective Midline Laparotomies After FAscia Closure Using Two Different Techniques of Running Sutures: COFACTOR-trial
Brief Title: Comparing Wound Complications After Elective Abdominal Surgery Using Two Closure Techniques
Acronym: COFACTOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Eman Sbaity, Instructor of Surgery, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIO-2017-038
Record Dates: First submitted 2018-04-24; First posted 2018-05-17 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-07

CONDITIONS: Wound Complication
Keywords: Incisional hernia; Wound infection; Midline laparotomy
MeSH Terms: conditions — Incisional Hernia; Wound Infection

STUDY DESIGN:
Intervention Model Description: 1:1 ratio
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard arm (No Intervention): In the standard arm, an average of one suture will be placed at each cm length of the wound, thus the number of sutures placed should be equal to the length of the wound in cm.
- Intervention arm (Experimental): The intervention arm will undergo the alternative/new closure technique with small and close fascia sutures, where each suture will be placed only 5 mm away from the fascia edge and 5 mm apart from the adjacent fascia suture.
  Interventions: Procedure: New closure technique

INTERVENTIONS:
Procedure: New closure technique — In the intervention arm, an average of two sutures will be placed at each cm length of the wound, thus the number of sutures placed should be equal to at least double the length of the wound in cm.The aim is to have a ratio of 4:1 between the overall lengths of the suture to the length of the wound being closed
  Other Names: Alternative closure technique
  Arms: Intervention arm

SUMMARY:
Wound complications, increased hospital stays and post-operative morbidity are all common following abdominal surgery. Abdominal closure complications are strongly associated with the closure technique and material used. The traditional closure technique used by surgeons is placing the wide and large stitches. A randomized controlled trial done in Sweden described a new closure technique in surgeries by placing the stitches closer to each other by using narrow. The results showed lower incidence of wound infections, hernias, and wound rupture. However, the study provides low quality evidence on the benefits of this new technique since it has numerous limitations like lack of standardization of suture size, lack of proper randomization, and heterogeneity in patient eligibility which will increase result bias. There is still a need for quality evidence on the effectiveness of this new closing technique procedure at decreasing wound complications after the operation.

In this trial the investigators will compare two techniques in the closure of abdominal wounds in patients undergoing abdominal surgery. The first technique will be the traditional closure technique currently used in abdominal surgery. The second technique will be using the new closure technique. The closure of abdominal wounds with small and close sutures using the new technique is expected to lower the incidence of hernia and wound complications as well as improve the quality of life of the patient. Potential candidates for the study are those who will be undergoing elective midline laparotomy at AUBMC. The patients and assessor of outcomes will be blinded and patients will be randomized to receive either the traditional or new closure operation technique. There are no anticipated risks for those participating in the study. All data and information collected will be kept confidential.

Hypothesis:

Closure of abdominal fascia in elective midline laparotomy incisions with small and close sutures compared to closure with conventional wide and distant sutures results in lower rates of wound rupture, incisional hernia, and wound infection, and improved quality of life.

Significance:

The results of this study will allow surgeons to assess the role of a new abdominal closure technique in decreasing short and long term postoperative complications, for a commonly performed procedure. This trial will generate evidence-based conclusions.

DETAILED DESCRIPTION:
Trial Design:

This trial is designed as a 1:1 randomized, controlled, patient and assessor-blinded, parallel design, superiority trial, with a primary endpoint of incisional hernia at one year.

Study Settings:

The investigators will conduct the study at the American University of Beirut Medical Center, which is an academic, tertiary referral center.

Prior to conducting this trial, the investigators will conduct a pilot study to study the feasibility of implementing the final trial by assessing items related to the institutional systems, the trial itself, and study subjects. The pilot study will assess the patient's response rate to participate in the trial, acceptance of patients to be examined daily by the research team, adherence of patients to the scheduled postoperative visits especially the one year follow up visit, and the proportion of loss to follow up. In the pilot, the investigators will also study the reliability of the randomization and allocation concealment strategy, and success of blinding of the research team from treatment allocation, efficacy of the training session and procedure video, consistency of evaluation among different surgeons performing the outcome assessments, and availability of the study team for the scheduled evaluations.

Strategies to improve adherence to intervention protocol:

The length of the fascia incision will be measured just before the surgeon starts the closure and this measurement will be documented by the research assistant (RA). After the wound is closed, the remaining suture length is measured again and documented. For a successful closure of the wound with this new technique, the utilized suture length should be 4 times the length of the wound. Approximately an additional 10 cm of suture length is needed to ensure proper tying of the knot after the conclusion of the suturing. The remaining suture length should reflect these two considerations. The circulating nurse will independently calculate the used and remaining suture length. The formula will be as follows: [Original Length of Suture (Length of suture remnants at the starting knot + Length of suture remnant at the finishing knot)]/ Length of the skin incision. If the final calculation result doesn't reflect the planned 4:1 ratio between the suture length and wound length, then the patient has to be removed from the study.

During the duration of hospital stay, it is the responsibility of the PI/study team to ensure proper and timely assessment of outcome measures. The study team will call the patients one week and 48 hours before the 30-day appointment and two weeks and one week before the one-year appointment to ensure show up

Relevant concomitant care and interventions during the trial:

Closure of the subcutaneous tissue and skin will be left at the discretion of the treating surgeon since currently there is no definitive evidence on the optimal methods following a laparotomy.

Whether to place drains or not in the subcutaneous tissue is also left to the discretion of the treating surgeon, since there is no consensus on this topic in the surgical literature.

Postoperative care of the patient during hospitalization and throughout the duration of the study will be performed according to usual care adopted by each surgeon.

Measures to prevent wound infections will be done following the hospital policy derived from the CDC guidelines on the prevention of surgical wound infections. Wound infection will be managed according to the general principles of skin opening and antibiotics.

Participant Timeline:

Enrollment:

After the primary attending introduces the study to the patients in the outpatient clinics or in the hospital during their admission period before surgery is performed, the RA will approach the patient and discuss the research study with them.

Assessments and Visits:

Daily visits to the participants will be conducted by the surgeon evaluator while in the hospital for the first 7 days to evaluate relevant outcome measures.

Two or three independent surgeon evaluators will be identified at our center to perform the clinical evaluation. The surgeon evaluator will be either a general surgeon or a vascular surgeon willing to dedicate time for the trial. She/he can't be the attending physician of the study subject. They will receive the training session with the remaining faculty who will enroll patients on the trial. Of note is that we elected to use physical examination as the method for abdominal incisional hernias detection because we are seldom interested in the clinically irrelevant hernias.

Sample Size:

In order to detect a drop of 12 % in the incidence of incisional hernia, with an alpha of 5% and 80% power, the investigators will need to recruit 114 patients in each arm and a total of 228 patients in the trial. The investigators are expecting a 30% loss to follow up, so our adjusted target recruitment will be 274 subjects in total.

Recruitment:

Possible candidates will be identified from surgery outpatient clinics during the preoperative visit. The attending surgeon will introduce briefly the trial to the patient, and if the patient agrees to participate, he will be approached by the RA. If a candidate was not approached in clinic, the RA will approach them prior to surgery, only after the attending physician gets the patient approval.

The expected recruitment rate is 2-3 patients per week. Consequently, it will take about two years to recruit a total of 274 patients. At AUBMC, the investigators currently perform 300 open laparotomies per 12 months. This recruitment rate will be tested in the pilot phase of the study.

Assignment of interventions

Sequence Generation:

Participants will be randomly assigned to their treatment in a 1:1 ratio, according to a computer generated schedule, stratified by type of surgery (vascular or non-vascular), using permuted blocks of variable sizes.

Allocation Concealment Mechanism:

Random sequence generation will be selected by an independent biostatistician, and the details of the blocking and block sizes will be saved in a separate document unavailable to those involved in the study including those enrolling patients, collecting data, evaluating outcomes, or analyzing data, so the investigators ensure concealment.

Data Collection Methods:

Data on basic demographics of the study subjects, relevant risk factors, confounders, and indication for laparotomy surgery will be collected at baseline using protocol-specific standardized case report forms, CRF. The CRF will be completed by the RA, following informed consent and prior to the surgical procedure. Data will be collected directly from the patient

Data Management:

The PI will perform spot checks on the data and will review weekly all the CRF and assessment collection sheets performed within each week.

The data will be stored on the American University of Beirut (AUB) intranet server and the CRFs will be stored in a locked cabinet by the PI for 3 years.

The investigators will provide a SOP (standard operating manual) detailing data management procedure to ensure consistency in case of change in the study members.

Statistical Methods:

The intervention arm (short and narrow stitches) will be compared to the standard arm (long and wide stitches) for the primary, secondary, and exploratory outcomes. The investigators will use the chi-square or Fischer exact test if the expected count of any of the outcomes is less than 5 per cell for analysis of incidence of dichotomous outcomes (fascia dehiscence, incisional hernia, wound seroma, wound infection, and intervention for wound complications). The investigators will use independent t-test for analysis of the continuous outcomes (pain score, and QOL measurement). The investigators will calculate relative risk with corresponding 95% confidence intervals to compare incidence of the dichotomous outcomes and The investigators will report difference in means for the continuous outcomes. SPSS version 20 will be used to conduct the analysis. A 2 sided p-value will be set at 5%.

Univariate analysis will be performed separately for the primary outcome and the two secondary outcomes. Univariate analysis will be conducted separately incisional hernia at one year ,intervention for wound complications at 30 day postoperative, and dehiscence at 30 days postoperative as the dependent variable and vascular indications, diabetes status, BMI, incision length, wound classification (clean, clean-contaminated, or contaminated) and operating surgeon as the independent variables. BMI will be categorized as normal, overweight, obese, and morbidly obese according to consensus BMI values cutoffs for these definitions. Wound status will be classified according to ACS wound classification system.

Multivariate analysis using logistic regression will be performed looking at how the primary outcome and each of the secondary outcome measures are affected by each of the above listed 4 covariates.

The investigators will perform subgroup analysis for the primary and secondary outcomes using chi-square according to the following variables: operation for vascular vs. non-vascular disease; obese vs. non-obese patients. The investigators anticipate that in the obese patients, the seroma and wound infections will be significantly less in the intervention versus the standard group. The investigators anticipate that the improvement in primary outcomes, especially in incidence of incisional hernia at one year will be more pronounced in the vascular surgeries.

The investigators will perform both intent-to-treat and per-protocol analysis for all outcome measures. The intent-to-treat analysis will include all patients in the arm to which they were randomized. Multiple imputation methods will be used to handle missing data. To assess the effect of missing data on the analysis, sensitivity analyses will be performed. The study biostatistician will perform best case scenario, worst case scenario, and group averages. For outcome measures missing from the 30 day assessment but available at discharge from the hospital, the biostatistician will use approach of "last observation carried further". The investigators will assess the baseline characteristics of those who will be lost to follow up, to help us understand what the potential outcomes were.

Data monitoring Committee (DMC):

The DMC committee will be independent of the principal investigator and the funders of the trial. It will be composed of a surgeon, internist, nurse, a biostatistician, and a representative from the patient advocacy office at AUB-MC.

The DMC will meet every other month, at times of scheduled interim analysis, and upon conclusion of the study.

Interim Analysis:

The interim analysis will be done using the O'Brien Fleming stopping rules 3 times throughout the study; upon recruiting quarter, two-quarters, and three-quarters of the study population.

Harms:

Any side effect will be reported and the subject will be managed according to the standard of care or the preference of the treating surgeon.

Ethics and Dissemination The investigators will submit this protocol, informed consent template, case report forms, and other study related appendices to the Institutional Review Board (IRB). The PI will submit progress reports to IRB annually till study termination.

Consent:

After the primary surgeon introduces the study to the patient, the RA will explain the study and invite the patients to sign the consent form. The subject will be given opportunity to ask questions about the study and will receive a copy of the consent forms signed by him/her.

Access to data:

At conclusion of the study, principal investigators and co-principal investigators will have full access to the identified data. Data will be handled respecting participants' confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Signed Informed Consent
* Undergoing an elective laparotomy through a midline incision
* Undergoing a midline laparoscopic procedure (midline laparoscopic extraction site)

Exclusion Criteria:

* Emergency surgery
* Laparotomy through an incision other than midline
* Previous midline laparotomy
* Presence of incisional or ventral hernia at time of laparotomy
* Incisional hernia repair
* Laparotomy surgery during pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia | 1 year
  We will define incisional hernia according to the European Society of Hernia: "any abdominal wall gap with or without bulge in the area of a postoperative scar perceptible or palpable by clinical examination or imaging". (7) Using both clinical exam and imaging if performed, these hernias will be described according to their location along the midline, size of the defect using vertical and transverse measurements, and reducibility of any protruding viscera upon lying down or following gentle pressure by the examining hand. Also, we will collect information whether the hernia is causing any pain, discomfort, decrease in mobility, or any incidence of incarceration where the hernia contents protrude and does not reduce to the abdomen upon gentle pressure.

SECONDARY OUTCOMES:
Fascial dehiscence or evisceration | 1 month postoperative
  Fascial dehiscence is defined as gapping of the fascia by at last 1 cm with loosening of the surgical sutures. This presents initially with increased serous fluid drainage from the wound. This may be self-limited or progress to a wider gap with herniation of the abdominal viscera, usually the small bowel or the greater omentum, through the defect. The excessive fluid drainage results in opening of the superficial skin incision in some patients and this necessitates emergency surgery for repeat closure of the abdominal wall.
Intervention rate for wound complications | 1 month postoperative
  Intervention includes incision and drainage for a wound infection, evacuation of a hematoma, aspiration of a seroma, or reoperation for a wound dehiscence.

OTHER OUTCOMES:
Wound seroma | 1 month postoperative
  Wound seroma defined as collection of serous fluid in the subcutaneous space, detected either clinically or by ultra-sound examination. o Wound seroma is an established risk factor for wound infection and further resultant morbidities
Wound infection | 1 month postoperative
  Wound infection will be defined according to the Centers of Disease Control CDC criteria for Surgical Site Infection SSI. Wound infection is a well known cause of fascia dehiscence. In addition, fascia closure technique resulting in fascia ischemia will result in deep surgical site infection, which in turn can lead to fascia dehiscence. The Sweden group believe that the wide fascia bite result in higher risk of fascia ischemia and thus delayed fascia healing or higher risk of deep wound (fascia) infection and higher risk of fascia gapping.
Intensity of Pain | up to 1 week
  Pain will be measured using "0-10 Numeric Pain Rating Scale" on post-operative day (POD) 1, POD 7, and on discharge (if the patient stays less than 7 days). The scale ranges from 0-10, 0 being the minimum score for pain intensity and 10 the maximum score for pain intensity. The values in the pain scale represent the pain level as follows: Zero means no pain at all, 1-3 means mild pain, 4-6 means moderate pain and 7-10 means severe pain.The research assistant will collect information on pain killers given to the patients post-operative. There are no sub scales in this measurement. This information will be taken into consideration when assessing pain intensity.
Quality of Life (QOL) | 1 year
  Quality of life will be measured using the "Short Form (SF-36) Health Survey Questionnaire", which has been validated in the Arabic language. The survey will assess the health related quality of life of the participants. The survey includes eight sections: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Aggregate scores are compiled as a percentage of the total points possible, using the Research ANd Development (RAND) scoring table. The scores from those questions that address each specific area of the functional health status are then averaged together, for a final score within each of the 8 sections measured. All 8 sections are scored in the same way.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Sbaity, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leaper DJ, van Goor H, Reilly J, Petrosillo N, Geiss HK, Torres AJ, Berger A. Surgical site infection - a European perspective of incidence and economic burden. Int Wound J. 2004 Dec;1(4):247-73. doi: 10.1111/j.1742-4801.2004.00067.x. PMID 16722874
- [Background] Bucknall TE, Cox PJ, Ellis H. Burst abdomen and incisional hernia: a prospective study of 1129 major laparotomies. Br Med J (Clin Res Ed). 1982 Mar 27;284(6320):931-3. doi: 10.1136/bmj.284.6320.931. PMID 6279229
- [Background] Wissing J, van Vroonhoven TJ, Schattenkerk ME, Veen HF, Ponsen RJ, Jeekel J. Fascia closure after midline laparotomy: results of a randomized trial. Br J Surg. 1987 Aug;74(8):738-41. doi: 10.1002/bjs.1800740831. PMID 3307992
- [Background] Rahbari NN, Knebel P, Diener MK, Seidlmayer C, Ridwelski K, Stoltzing H, Seiler CM. Current practice of abdominal wall closure in elective surgery - Is there any consensus? BMC Surg. 2009 May 15;9:8. doi: 10.1186/1471-2482-9-8. PMID 19442311
- [Background] Diener MK, Voss S, Jensen K, Buchler MW, Seiler CM. Elective midline laparotomy closure: the INLINE systematic review and meta-analysis. Ann Surg. 2010 May;251(5):843-56. doi: 10.1097/SLA.0b013e3181d973e4. PMID 20395846
- [Background] Millbourn D, Cengiz Y, Israelsson LA. Effect of stitch length on wound complications after closure of midline incisions: a randomized controlled trial. Arch Surg. 2009 Nov;144(11):1056-9. doi: 10.1001/archsurg.2009.189. PMID 19917943
- [Background] Muysoms FE, Miserez M, Berrevoet F, Campanelli G, Champault GG, Chelala E, Dietz UA, Eker HH, El Nakadi I, Hauters P, Hidalgo Pascual M, Hoeferlin A, Klinge U, Montgomery A, Simmermacher RK, Simons MP, Smietanski M, Sommeling C, Tollens T, Vierendeels T, Kingsnorth A. Classification of primary and incisional abdominal wall hernias. Hernia. 2009 Aug;13(4):407-14. doi: 10.1007/s10029-009-0518-x. Epub 2009 Jun 3. PMID 19495920
- [Derived] El Charif MH, Hassan Z, Hoballah J, Khalife M, Sbaity E. Protocol for a randomized controlled trial comparing wound COmplications in elective midline laparotomies after FAscia Closure using two different Techniques Of Running sutures: COFACTOR trial. Trials. 2020 Jul 2;21(1):608. doi: 10.1186/s13063-020-04507-8. PMID 32616017